CLINICAL TRIAL: NCT03364868
Title: Oral Insulin Therapy for Prevention of Autoimmune Diabetes
Brief Title: GPPAD-POInT (Global Platform of Autoimmune Diabetes - Primary Oral Insulin Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Helmholtz Zentrum München (Industry); University Hospital Carl Gustav Carus (Other); Kinderkrankenhaus auf der Bult (Other); Skane University Hospital (Other); Universitaire Ziekenhuizen KU Leuven (Other); Medical University of Warsaw (Other); University of Oxford, Clinical Vaccine Research and Immunisation Education (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GPPAD-03-POInT
Record Dates: First submitted 2017-11-13; First posted 2017-12-07 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; T1D; diabetes mellitus; oral insulin; oral tolerance; autoantigen; self tolerance; prevention; at risk for developing type 1 diabetes; juvenile diabetes; autoimmune diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral insulin capsule (dose escalation using 3 dose strengths) (Experimental): Dose 1 is 7.5 mg rH-insulin crystals; dose 2 is 22.5 mg rH-insulin crystals; dose 3 is 67.5 mg rH-insulin crystals. The insulin crystals are formulated together with filling substance (microcrystalline cellulose to a total weight of 200 mg) and contained in hard gelatine capsules. The study treatment will be given orally.
  Interventions: Drug: Oral Insulin
- Placebo capsule (Placebo Comparator): Daily treatment with placebo capsules containing filling substance (microcrystalline cellulose).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oral Insulin — treatment starting at 4 months - 7 months until age 3.0 years; dose escalation scheme: daily treatment with 7.5 mg or placebo for 2 months; increasing to daily treatment with 22.5 mg or placebo for the following 2 months; increasing to daily treatment with 67.5 mg or placebo until the end of the treatment period.
  Arms: oral insulin capsule (dose escalation using 3 dose strengths)
Other: Placebo — treatment starting at age 4 months - 7 months until age 3.0 years; daily treatment with insulin or placebo capsules containing filling substance (microcrystalline cellulose).
  Arms: Placebo capsule

SUMMARY:
The GPPAD-POInT Study is designed as a randomized, placebo-controlled, double blind, multicentre, multinational primary prevention phase IIb study aiming to induce immune tolerance to beta-cell autoantigens through regular exposure to oral insulin for a period of 29 to 32 months. The hypothesis is that regular exposure to oral insulin throughout the period in life where beta-cell autoimmunity usually initiates will tolerize against insulin and train the body's immune system to recognize the treatment product without reacting adversely to it in a manner seen in children who develop T1D. This immune tolerance induction therapy would reduce the likelihood of beta-cell autoimmunity. The study objective is to determine whether daily administration of oral insulin from age 4 months - 7 months until age 3.00 years to children with elevated genetic risk for type 1 diabetes reduces the cumulative incidence of beta-cell autoantibodies and diabetes in childhood.

DETAILED DESCRIPTION:
The GPPAD-POInT-Study aims to determine whether daily administration of oral insulin to children from age 4 months - 7 months with elevated genetic risk for type 1 diabetes reduces the cumulative incidence of beta-cell autoantibodies and diabetes in childhood. The purpose of the GPPAD-POInT-Study is to induce immune tolerance to beta-cell autoantigens through regular exposure to oral insulin for a period of 29 to 32 months. Together with the results of the Pre-POINT-Early Study, this phase IIb study aims to investigate and consolidate the findings from the pilot Pre-POINT Study, namely safety and immune efficacy at a daily dose of 67.5 mg oral insulin. Since babies and young children will be tested in the GPPAD-POInT-Study, the 67.5 mg dose will be reached by dose escalation starting at 7.5 mg for 2 months, followed by exposure to 22.5 mg for 2 months, and reaching the desired 67.5 mg dose. The GPPAD-POInT-Study aims to recruit 1040 children into the trial.

The active substance for oral application is human insulin. Oral Insulin will be applied as a capsule containing 7.5, 22.5 and 67.5 mg of the active substance together with filling substance microcrystalline cellulose.

ELIGIBILITY:
Inclusion Criteria:

1. Infant between the ages of 4 months and 7 months at the time of randomization.

2. A high genetic risk (>10%) to develop beta-cell autoantibodies by age 6 years:

1. For infants without a first degree family history of type 1 diabetes, high genetic risk is defined as a DR3/DR4-DQ8 or DR4-DQ8/DR4-DQ8 genotype, and a genetic risk score that is >14.4.
2. For infants with a first degree family history of type 1 diabetes, high genetic risk is defined as having HLA DR4 and DQ8, and none of the following protective alleles: DRB1*1501, DQB1*0503.
3. Solid foods introduced into diet of infant
4. Written informed consent signed by the custodial parent(s).

Exclusion Criteria:

1. Concomitant disease or treatment that may interfere with the assessments, as judged by the investigators.
2. Any condition that could be associated with poor compliance.
3. Any medical condition or medical condition coexisting, which, in the opinion of the investigator, may jeopardize the participant's safe participation in the study.
4. Diagnosis of diabetes at the time of recruitment.
5. Participation in another clinical trial.

Ages: 4 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1050 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
The development of persistent confirmed multiple beta-cell autoantibodies | elapsed time from treatment assignment (baseline) to first positive sample visit (>2 beta-cell antibodies) in children who develop persistent confirmed multiple beta-cell antibodies. Primary outcome can develop any time up to last study visit at 7.5 yrs
  development of persistent confirmed multiple beta-cell autoantibodies (defined as confirmed IAA, confirmed GADA, confirmed IA-2A, or confirmed ZnT8A in two consecutive samples, AND a confirmed second antibody from these four antibodies in one sample.
The development of diabetes | elapsed time from random treatment assignment (baseline) to the development diabetes (date of diagnosis). This primary outcome measure can develop any time during treatment or follow-up period up to the last study visit at 7.5 years of age
  OGTT criteria or clinical criteria for diabetes as defined by the American Diabetes Association (ADA).

SECONDARY OUTCOMES:
Any persistent confirmed beta-cell autoantibody or diabetes | elapsed time from treatm. assignm. (baseline) to 1st pos. sample for >1 beta-cell antibody in children who developed persist. confirm. beta-cell antibodies OR diabetes onset, whichever is first. outcome can develop any time up to last visit at 7.5 yr
  At least one confirmed autoantibody, in two consecutive samples, including GADA, IA-2A, IAA, ZnT8A, or TS7A, or diabetes as defined by the American Diabetes Association (ADA).
Persistent confirmed IAA. | elapsed time from treatment assignment (baseline) to first sample that is positive for IAA in children who develop persistent confirmed IAA. Outcome can develop any time during treatment or follow-up period up to the last study visit at 7.5 years of age.
  Confirmed IAA in two consecutive samples.
Persistent confirmed GADA. | elapsed time from treatment assignment (baseline) to the first sample that is positive for GADA in children who develop persistent confirmed GADA. Outcome can develop any time up to the last study visit at 7.5 years of age
  Confirmed GADA in two consecutive samples.
Abnormal glucose tolerance (AGT) defined by dysglycemia or diabetes. | elapsed time from treatment assignment to the date at which abnormal glucose tolerance or diabetes is diagnosed. Outcome can develop any time up to the last study visit at 7.5 years of age
  Dysglycemia is defined as impaired fasting plasma glucose of ≥110 mg/dL (6.1 mmol/L), or impaired 2-hour glucose of ≥140 mg/dL (7.8 mmol/L), or high glucose levels at intermediate time points on OGTT (30, 60, 90 min) levels of ≥200mg/dL (11.1 mmol/L)). Diabetes is defined according to the criteria of the American Diabetes Association (ADA).

CONTACTS AND LOCATIONS:
Locations (7):
- University Hospitals Leuven, Faculty of Medicine, Catholic University of Leuven, Leuven, Belgium, Leuven, Belgium
- Germany (3):
  - Forschergruppe Diabetes, Klinikum rechts der Isar, Technische Universität München, Munich, Germany, Munich, Bavaria
  - AUF DER BULT, Kinder- und Jugendkrankenhaus, Hanover, Germany, Hanover, Lower Saxony
  - Klinik und Poliklinik f. Kinder und Jugendmedizin, Universitätsklinikum Carl Gustav Carus, Technische Universität Dresden, CRTD/DFG-Forschungszentrum für Regenerative Therapien, Dresden, Germany, Dresden, Saxony
- Medical University of Warsaw, Department of Paediatrics, Warsaw, Poland, Warsaw, Poland
- Lund University Dep. of Clinical Sciences Malmo, Skane University Hospital SUS, University Hospital MAS, Malmo, Sweden, Malmo, Sweden
- Department of Paediatrics Clinical Vaccine Research and Immunisation Education, Children's Hospital, Headington, Oxford, UK, Oxford, United Kingdom

REFERENCES:
- [Derived] Ziegler AG, Achenbach P, Weiss A, Berner R, Casteels K, Elding Larsson H, Haupt F, Hommel A, Jacobs A, Kordonouri O, Lundgren M, Oltarzewski M, Pfirrmann M, Snape MD, Szypowska A, Todd JA, Vatish M, von dem Berge T, Winkler C, Bonifacio E; GPPAD-POInT Study Group. Efficacy of once-daily, high-dose, oral insulin immunotherapy in children genetically at risk for type 1 diabetes (POInT): a European, randomised, placebo-controlled, primary prevention trial. Lancet. 2025 Nov 29;406(10519):2564-2576. doi: 10.1016/S0140-6736(25)01726-X. Epub 2025 Nov 11. PMID 41237794
- [Derived] Jacobsen LM, Schatz DA. Insulin immunotherapy for pretype 1 diabetes. Curr Opin Endocrinol Diabetes Obes. 2021 Aug 1;28(4):390-396. doi: 10.1097/MED.0000000000000648. PMID 34091488
- [Derived] Ziegler AG, Achenbach P, Berner R, Casteels K, Danne T, Gundert M, Hasford J, Hoffmann VS, Kordonouri O, Lange K, Elding Larsson H, Lundgren M, Snape MD, Szypowska A, Todd JA, Bonifacio E; GPPAD Study group. Oral insulin therapy for primary prevention of type 1 diabetes in infants with high genetic risk: the GPPAD-POInT (global platform for the prevention of autoimmune diabetes primary oral insulin trial) study protocol. BMJ Open. 2019 Jun 28;9(6):e028578. doi: 10.1136/bmjopen-2018-028578. PMID 31256036